CLINICAL TRIAL: NCT05848674
Title: CABIN (CArdiac Brief INtervention): A Feasibility Study to Promote Engagement With Cardiac Rehabilitation Through an Early, Personalised, Holistic Intervention
Brief Title: CArdiac Brief INtervention: A Feasibility Study to Promote Engagement With Cardiac Rehabilitation
Acronym: CABIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other); South Eastern Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Gareth Thomson, Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B23/01
Record Dates: First submitted 2023-04-17; First posted 2023-05-08 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Group 1: Intervention; Group 2: Control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): CABIN will be delivered in a single session to each participant (one-to-one) of the intervention group by a Research Assistant who is a cardiac nurse with over 20 years of clinical experience in cardiac rehabilitation. A private space at a Coronary Care Unit (Royal Victoria Hospital or Ulster Hospital) will be used for intervention delivery before patient discharge. Intervention delivery should take approximately 20 minutes.
  Interventions: Other: CArdiac Brief INtervention (CABIN)
- Control Group (Other): A Research Fellow will deliver (one-to-one) a refined version of CABIN prior to patient discharge from a Coronary Care Unit (Royal Victoria Hospital or Ulster Hospital). A private space will be used, with delivery taking approximately 10 minutes.
  Interventions: Other: Refined version of CABIN

INTERVENTIONS:
Other: CArdiac Brief INtervention (CABIN) — CABIN is designed as a brief intervention with a facilitated discussion between a patient and a nurse, with the provision of a short leaflet that summarises information and acts as an aide memoir. The discussion takes place in a quiet area and is intended to last 15-20 minutes. CABIN involves a nurse listening to the patient and recognising any concerns he / she may have and / or identifying erroneous beliefs. It also provides the patient with personalised education on coronary artery disease and cardiac rehabilitation (i.e., information about stenting, stent placement, medication, and purpose / potential benefits of cardiac rehabilitation), along with facilitating psychological and emotional support discussions with a nurse (i.e., explaining causes of a STEMI, discussing support / treatment options, and exploring methods of improving health).
  Arms: Intervention Group
Other: Refined version of CABIN — Participants of the control group will receive a refined version of CABIN, which excludes psychological and emotional support discussions with a nurse and details some standard discharge information (information about coronary artery disease and stenting / stent placement).
  Arms: Control Group

SUMMARY:
Background:

An ST-elevation myocardial infarction (STEMI) is a specific type of heart attack. In a previous study, patients requested more mental and emotional support after a STEMI. To provide this support, the research team worked with hospital staff and patients to create a brief intervention called CABIN (CArdiac Brief INtervention), which involves a short discussion between a patient and a nurse, along with a leaflet that summarises the information discussed.

Aim:

To test if the plan for giving CABIN to patients after a STEMI is suitable, and to explore what impact the intervention may have on mental and emotional well-being, along with knowledge about their condition.

Methods:

Forty patients who had a STEMI will be recruited from two hospital centres in Northern Ireland (Royal Victoria Hospital and Ulster Hospital). Participants will be randomly put in a group who receive the full CABIN intervention or a group who receive a shortened version of CABIN. Both groups will receive their respective interventions before leaving the hospital, which will take about twenty minutes. Participants will be asked to complete brief questionnaires before the intervention, after the intervention, 3-4 weeks from diagnosis, and 14 weeks from diagnosis. At the end of the study, patients who took part and staff from the hospitals will be asked to complete an exit interview (patients) or a focus group (staff), which will provide information about their experience of the study / intervention and changes required.

Outcome of Study:

If the study is suitable for patients and appropriate for staff to deliver, the research team will examine the effectiveness of CABIN in a larger study, which may lead to the intervention being used in clinical practice to improve cardiac rehabilitation uptake and outcomes for patients after a STEMI.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over.
* Confirmed diagnosis of STEMI.
* Physically and mentally capable of participation (judged by Cardiologist or Nurse).
* Willing to provide informed consent.

Exclusion Criteria:

* Lacking capacity to give consent (judged by Cardiologist or Nurse).
* Under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
The percentage of eligible patients who agreed to participate in the study. | Through study completion, an average of 1 year.
  The measurement of recruitment rate will allow the efficiency of the recruitment strategy to be assessed, with this information enabling the identification of potential issues and informing the required duration of the recruitment period for a larger study.
The percentage of intervention delivered (Dose) | Week 1
  Dose will assess the completeness of intervention delivery, which will inform the feasibility of CABIN implementation. This information will be collected via an intervention checklist that is completed by the Research Assistant following each intervention session.
The percentage of recruited participants providing data for each baseline and outcome measure. | Through study completion, an average of 1 year.
  The completeness of baseline and outcome measures will be determined as missing data may jeopardise the power of a future study. The Research Fellow will record details about data collection in the study log, which will highlight any problems or required changes to improve data collection for a future study.
Perspectives of patients on research design and intervention delivery. | Week 14
  Participants will be invited to a semi-structured interview upon study completion to discuss:
  1. Acceptability of intervention (i.e., issues for development, required corrections, additional areas for inclusion, aspects enjoyed by participants, and barriers and facilitators to participation).
  2. Context (i.e., factors influencing study / intervention delivery and functioning, for instance, time and resources).
  3. Possible mechanisms of impact (i.e., exploring how intervention activities may trigger change for participants).
Perspectives of clinical staff on research design and intervention delivery. | Week 14
  Coronary care unit and cardiac rehabilitation staff will be invited to focus groups to discuss:
  1. Acceptability of intervention (i.e., issues for development, required corrections, additional areas for inclusion, aspects enjoyed by participants, and barriers and facilitators to participation).
  2. Context (i.e., factors influencing study / intervention delivery and functioning, for instance, time and resources).
  3. Possible mechanisms of impact (i.e., exploring how intervention activities may trigger change for participants).

SECONDARY OUTCOMES:
Change from baseline in Coronary Artery Disease Education Questionnaire, Short Version (CADE-Q SV) score | Baseline, Week 1, Week 4, and Week 14.
  CADE-Q SV evaluates patients' knowledge of coronary artery disease and core components of cardiac rehabilitation. Score will be reported as the number of 20 questions answered correctly. A higher score represents a better outcome.
  Change = (follow-up measurement score - baseline score).
Change from baseline in Brief Illness Perception Questionnaire score | Baseline, Week 1, Week 4, and Week 14.
  Brief Illness Perception Questionnaire rapidly assesses the cognitive and emotional representations of illness. Scored on a 10-point Likert scale across eight domains.
  Change = (follow-up measurement score - baseline score).
Change from baseline in the Hospital Anxiety and Depression Scale score. | Baseline, Week 1, Week 4, and Week 14.
  The Hospital Anxiety and Depression Scale measures states of depression and anxiety. Each question is scored between zero (no impairment) and three (severe impairment), with a maximum score of 21 for anxiety or depression.
  Change = (follow-up measurement score - baseline score).
Change from baseline in Personal Wellbeing Score | Baseline, Week 1, Week 4, and Week 14.
  Personal Wellbeing Score measures health status and health confidence. Each item is scored as follows: Disagree=0, Neutral=1, Agree=2 and Strongly Agree=3. A high score is better than a low score.
  Change = (follow-up measurement score - baseline score).
Number of cardiac rehabilitation sessions attended. | Week 14.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Fitzsimons, PhD, Principal Investigator — Queen's University, Belfast; Judy Bradley, PhD, Principal Investigator — Queen's University, Belfast
Locations (2):
- United Kingdom (2):
  - Royal Victoria Hospital, Belfast Health and Social Care Trust, Belfast, Antrim
  - Ulster Hospital, South Eastern Health and Social Care Trust, Dundonald, Down

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson G, Caughers G, Bradley J, Donnelly P, Mooney M, Fitzsimons D. The feasibility of delivering cardiac brief intervention to patients following ST-elevation myocardial infarction: Protocol for a pilot randomised controlled trial. PLoS One. 2024 Jul 2;19(7):e0306406. doi: 10.1371/journal.pone.0306406. eCollection 2024. PMID 38954674